CLINICAL TRIAL: NCT03886233
Title: Treatment Outcome of Uveitis in Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elham youssif Ahmed Ali, Assiut, Assiut University
Other Study IDs: IRB000188
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Autoimmune Uveitis
MeSH Terms: interventions — Biological Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional Treatment for Autoimmune uveitis: Corticosteroids are considered the gold standard in management of acute AU. They can only be administered after excluding infectious origin. Their use for prolonged time and/ or in high doses may be associated with serious adverse events . Therefore, it is necessary to combine them with other immunosuppressive drugs.Based on their mechanism of action, immunosuppressives are divided into alkylating agents (cyclophosphamide and chlorambucil), antimetabolites (methotrexate, azathioprine, and Mycophenolate Mofetil), and calcineurin inhibitors (cyclosporine, tacrolimus and sirolimus).Dosage form, dosage, frequency and duration differ according to age and case severity.
  Interventions: Drug: Corticosteroid Series
- Biological Treatment for Autoimmune uveitis: Biological anti-inflammatory agents (for exapmle antagonists of tumor necrosis factor alpha like Infliximab and adalimumab) are also showing very promising results. In many cases, these agents will be seen listed as first choice in some autoimmune diseases, depending on the patient's history, age, sex, type and severity of the inflammatory disease.

INTERVENTIONS:
Drug: Corticosteroid Series — immunosuppressives are divided into alkylating agents (cyclophosphamide and chlorambucil), antimetabolites (methotrexate, azathioprine, and Mycophenolate Mofetil), and calcineurin inhibitors (cyclosporine, tacrolimus and sirolimus) Biological anti-inflammatory agents (for exapmle antagonists of tumor necrosis factor alpha like Infliximab and adalimumab).
  Other Names: Immunosuppressive drugs; Biological therapy
  Groups: Traditional Treatment for Autoimmune uveitis

SUMMARY:
reviewing the outcomes of patients with uveitis caused by autoimmune diseases treated at Assiut University Hospital at the Ophthalmology and Rheumatology and Rehabilitation Departments.

DETAILED DESCRIPTION:
Autoimmune uveitis (AU) is an inflammation of the uvea caused by either an autoimmune reaction to self-antigens or an innate inflammatory reaction secondary to an external stimulus. Corticosteroids are considered the gold standard in management of acute AU, but it is necessary to combine them with other immunosuppressive drugs. Finally, biological anti-inflammatory agents (for exapmle antagonists of tumor necrosis factor alpha like Infliximab and adalimumab) are also showing very promising results. Follow-up visits of subjects with uveitis must be frequent and focused on monitoring the recurrence of acute outbreaks, , if any. They should be aimed to determine the evolution of inflammatory signs until their complete resolution, thus ensuring the least possible consequences. After the initial phase of the treatment, the duration of use of the maintenance medication is directly related to the diagnosis, treatment and control of the underlying disease. This will help to determine if a patient is badly controlled and requires a more aggressive therapeutic plan. Also, a complete physical exam must be done each time the patient sees to the physician in order to monitor ophthalmological complications or development of adverse effects secondary to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Uveitis with clinical features of autoimmune disease;

Exclusion Criteria:

* Other infectious and non-infectious uveitic etiologies that may mimic the given clinical presentation of autoimmune uveitis;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include uveitis caused by autoimmune diseases. Uveitis can be anterior (including iritis or iridocyclitis). Intermediate uveitis or vitritis involves the vitreous cavity and may involve the pars plana. Finally, posterior uveitis is divided in three types: choroiditis, retinochoroiditis, and chorioretinitis. In diffuse involvement or when uveitis affects many areas, it is described as panuveitis.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
determination the best method for treatment of autoimmune uveitis | 2 years
  compare the rates of treatment failure in the management of autoimmune uveitis between patients who received steroids, immunosuppressive drugs or biological therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan L Fahmy, Prof., Study Chair — Assiut University; Mohamed G Saleh, lecturer, Study Director — Assiut University